CLINICAL TRIAL: NCT05699681
Title: Correlation of Right Atrial Strain With Pulmonary Hypertension, Right Ventricular Function And Outcome In Pediatric Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Subhrashis Guha Niyogi, Principal Investigator, Division of Cardiac Anaesthesia, Department of Anaesthesia and Intensive Care, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: NK/6412/Study/494
Record Dates: First submitted 2022-12-12; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Children aged below 12 years undergoing elective cardiac surgery for congenital heart disease with left to right shunt with prior evidence of pulmonary arterial hypertension on preoperative echocardiography
  Interventions: Diagnostic Test: Transthoracic and transesophageal echocardiography

INTERVENTIONS:
Diagnostic Test: Transthoracic and transesophageal echocardiography — After induction of anaesthesia and stabilization of hemodynamics, transthoracic echocardiography will be done on a GE Vivid e9 workstation (GE Vingmed, Horton, Norway) with MS5 transthoracic probe with synchronized ECG.
  From TTE the following views and measurements will be acquired :
  * Apical four chamber (A4C) view
  * Apical two chamber view (A2C) view
  * Right ventricle (RV) focused A4C view
  * Right ventricular systolic pressure (RVSP)
  * Pulmonary arterial acceleration time (PAAT),
  * Tricuspid annular plane systolic excursion (TAPSE),
  * Tricuspid annular plane systolic velocity (s'),
  * Right ventricular fractional area change (RV FAC)
  * RV free wall strain,
  * RV myocardial performance index (MPI),
  * RV isovolumic relaxation time (IVRT),
  * RV isovolumic acceleration time (IVA)
  Invasive PA pressure measurement will be done after surgical exposure with a fine needle and a zeroed transducer by the Surgeon.
  Other Names: Measurement of Pulmonary arterial pressure

SUMMARY:
This observational study aims to assess correlation of right atrial strain measured by two-dimensional speckle tracking echocardiography with intraoperatively measured pulmonary artery pressures, other indices of right ventricular function and short term postoperative outcome.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective cardiac surgery for congenital heart disease with left to right shunt
* Prior evidence of pulmonary arterial hypertension on preoperative echocardiography.

Exclusion Criteria:

* Neonates
* Children with history of previous cardiac surgery,
* Hemodynamic instability
* Non-sinus rhythm

Ages: 1 Month to 12 Years | Sex: All
Age Groups: Child
Study Population: As described above.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Correlation of right atrial strain measured by two-dimensional speckle tracking echocardiography with intraoperatively measured systolic pulmonary artery pressures. | For RA strain : after induction of anesthesia, before CPB institution. For pulmonary artery pressures, after induction of anesthesia, before CPB institution, and 10 min after separation from CPB, before sternal closure.
  RA strain estimation will be done from the TTE images in RV focused A4C view, tracing the endocardial border from tricuspid annulus to tricuspid annulus along RA lateral wall to roof to septal wall.
  After optimizing the region of interest and automated speckle tracking for longitudinal strain and the following parameters will be measured :
  * RA reservoir strain : difference of the strain value at tricuspid valve opening minus ventricular end-diastole (positive value).
  * RA conduit strain : difference of the strain value at the onset of atrial contraction minus tricuspid valve opening (negative value).
  * RA contractile strain : difference of the strain value at ventricular end- diastole minus onset of atrial contraction (negative value).

SECONDARY OUTCOMES:
Correlation of right atrial strain measured by two-dimensional speckle tracking echocardiography with other indices of right ventricular function. | For RA strain and RV function : after induction of anesthesia, before CPB institution.
  From TTE the following views and measurements will be acquired :
  Apical four chamber (A4C) view Apical two chamber view (A2C) view Right ventricle (RV) focused A4C view Right ventricular systolic pressure (RVSP) Pulmonary arterial acceleration time (PAAT), Tricuspid annular plane systolic excursion (TAPSE), Tricuspid annular plane systolic velocity (s'), Right ventricular fractional area change (RV FAC) RV free wall strain, RV myocardial performance index (MPI), RV isovolumic relaxation time (IVRT), RV isovolumic acceleration time (IVA)
Correlation of right atrial strain measured by two-dimensional speckle tracking echocardiography with short term postoperative outcome as defined by duration of mechanical ventilation and duration of ICU stay. | Preoperative (post induction, pre-CPB) RA reservoir, conduit and contractile strain will be correlated with duration of mechanical ventilation, and duration of ICU stay, measured on 30 days post-operative follow up.
  Duration of mechanical ventilation will be measured from time of shifting out from the operating room to first extubation. Similarly, ICU stay will be measured from the date of surgery to shifting to general ward.

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Institute of Medical Education & Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No